CLINICAL TRIAL: NCT01744262
Title: A Comparison of Totally Intravenous and Inhalation Anesthesia for Intraocular Pressure During Robot-Assisted Laparoscopic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2011-0034
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Prostate Cancer
Keywords: intraocular pressure, total intravenous anesthesia, laparoscopic prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Anesthesia, Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhalational anesthesia group (Active Comparator)
  Interventions: Drug: Inhalation Anesthesia
- Total intravenous anesthesia group (Experimental)
  Interventions: Drug: Total intravenous anesthesia

INTERVENTIONS:
Drug: Total intravenous anesthesia — Anesthesia induction with intravenous propofol (effect site concentration 2.5 µg/mL) and remifentanil (effect site concentration 3 ng/mL) using target controlled infusion (TCI). Anesthesia maintenance with propofol effect site concentration 1.5~4 µg/mL and remifentanil effect site concentration 2~5 ng/mL.
  Arms: Total intravenous anesthesia group
Drug: Inhalation Anesthesia — Anesthesia induction with intravenous propofol bolus of 1.5~2.5 mg/kg and remifentanil (effect site concentration 3 ng/mL)using target controlled infusion (TCI). Anesthesia maintenance with sevoflurane 1.5~2.0 % and remifentanil effect site concentration 2~5 ng/mL.
  Arms: Inhalational anesthesia group

SUMMARY:
Robot-assisted laparoscopic radical prostatectomy (RALRP) has gained popularity during the past decade and has widely replaced conventional open prostatectomy in many institutions due to reduced blood loss, nerve sparing, less postoperative pain and shorter hospital stay. However, laparoscopic surgery is performed with intraperitoneal carbon dioxide insufflation, which leads to increased intraocular pressure (IOP). In particular, robot-assisted laparoscopic radical prostatectomy (RALRP) usually requires a steep Trendelenburg position and often prolonged insufflation times, which is known to effect the increase in IOP during surgery and may result in ophthalmic complications such as postoperative vision loss (POVL). The majority of patients undergoing RALRP is old aged and often present with comorbidities. Advanced age, underlying diabetes mellitus (DM) or hypertension renders the patient vulnerable to damage due to increased IOP. Moreover, the possibility of the patient having undiagnosed glaucoma is also increased, and therefore methods to prevent such complications are needed. As of now, intravenous hypnotic agents, inhalation anesthetics and opioids have been reported to decrease IOP by relaxing extraocular muscle tone and increasing aqueous humour outflow to some extent. Among these agents, propofol has been reported to be more effective than other inhalational anesthetics in decreasing IOP. The goal of this prospective, randomized controlled trial is to compare the effect of propofol and sevoflurane on IOP in patients undergoing RALRP in the steep Trendelenburg position with carbon dioxide pneumoperitoneum.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class 1 or 2
2. Adults over the age of 20 and under 70
3. Patients undergoing robot-assisted laparoscopic radical prostatectomy
4. Patients that have given informed consent

Exclusion Criteria:

1. Patients with known ophthalmic diseases (glaucoma, diabetic retinopathy, cataract, retinal detachment)
2. Patients with history of ophthalmic surgery
3. Patients with high baseline intraocular pressure (over 30 mmHg)
4. Patients with active cardiac conditions (unstable angina, congestive heart failure)
5. Patients with uncontrolled hypertension (diastolic blood pressure > 110 mmHg)
6. Patients with history of allergic reactions to propofol
7. Illiterate patients

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Changes in intraocular pressure during pneumoperitoneum in the steep Trendelenburg position
  Before induction of anesthesia (T0), 5 minutes after induction of anesthesia (T1), 5 minutes after pneumoperitoneum (T2), 30 minutes after steep Trendelenburg position with pneumoperitoneum (T3), 5 minutes after returning to horizontal position with pneumoperitoneum (T4), 5 minutes after desufflation (T5), 5 minutes after awakening in the operating room (T6), 60 minutes after awakening in the recovery room (T7), 24 hours after the operation (T9)

REFERENCES:
- [Derived] Yoo YC, Shin S, Choi EK, Kim CY, Choi YD, Bai SJ. Increase in intraocular pressure is less with propofol than with sevoflurane during laparoscopic surgery in the steep Trendelenburg position. Can J Anaesth. 2014 Apr;61(4):322-9. doi: 10.1007/s12630-014-0112-2. Epub 2014 Feb 4. PMID 24500661